CLINICAL TRIAL: NCT02394418
Title: Comparison of Sedative Effects of Sevoflurane, Propofol and Dexmedetomidine on the Clinical Course of Delirium and Neuroinflammation in Mechanically Ventilated Patients
Brief Title: Effect of Sevoflurane, Propofol and Dexmedetomidine on Delirium & Neuroinflammation in Mechanically Ventilated Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: for technical reasons
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Valery V. Likhvantsev, Professor, senior researcher, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-D-P-MV-220115
Record Dates: First submitted 2015-01-27; First posted 2015-03-20 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Sevoflurane; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sevoflurane (Active Comparator): Treatment of delirium by inhaled sevoflurane
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Treatment of delirium by propofol i.v. infusion
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Treatment of delirium by dexmedetomidine i.v. infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Sevoflurane — Treatment of delirium by inhaled sevoflurane
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Propofol — Treatment of delirium by propofol i.v. infusion
  Other Names: Diprivan
  Arms: Propofol
Drug: Dexmedetomidine — Treatment of delirium by dexmedetomidine i.v. infusion
  Other Names: Dexdor
  Arms: Dexmedetomidine

SUMMARY:
Assessment of sedative effects of sevoflurane, dexmedetomidine and propofol on the clinical course of delirium, SIRS and neuroinflammation in mechanically ventilated patients using CAM-ICU scale, GSK-3beta and protein S100b in serum.

ELIGIBILITY:
Inclusion Criteria:

* presence of delirium

Exclusion Criteria:

* presence of Alzheimer's disease
* any mental disorder
* presence of cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Duration of Delirium | up to 5 days
  Delirium assessment by CAM-ICU scale

SECONDARY OUTCOMES:
Change of protein S100b in serum | from delirium onset up to 5 days
Change of GSK-3beta in serum | from delirium onset up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, MD,PhD, Principal Investigator — Moscow Regional Research Clinical Institute